CLINICAL TRIAL: NCT04201236
Title: Comparison of the Effectiveness of Inspiratory Muscle Training and Oropharyngeal Exercises in Patients With Obstructive Sleep Apnea Syndrome: a Randomized Controlled Trial
Brief Title: Oropharyngeal Exercises and Inspiratory Muscle Training in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, NUREL ERTURK, Principal Investigator, Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/11
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; oropharyngeal exercises; inspiratory muscle training; sleep quality
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oropharyngeal exercises (Experimental): Oropharyngeal exercises include soft palate, tongue and facial muscle exercises as well as stomatognathic function exercises. Training sessions were held once a day, 5 days a week for 12 weeks under the supervision of a mirror.
  Interventions: Other: oropharyngeal muscles strengthening exercise
- Inspiratory muscle training (Experimental): The inspiratory muscle training group was administered for 12 weeks starting from 30% of maximal oral pressure, 7 days a week, 15 minutes twice a day. Patients came to the control once a week, mouth pressures were measured and training pressure was adjusted in 30% of the new value.
  Interventions: Other: respiratory muscle strengthening exercise
- Control (No Intervention): This group was only monitorized without any rehabilitation intervention.

INTERVENTIONS:
Other: respiratory muscle strengthening exercise — These exercises strengthen locally inspiratory muscles. IMT can be done with threshold loaded devices.
  Arms: Inspiratory muscle training
Other: oropharyngeal muscles strengthening exercise — These exercises strengthen locally oropharyngeal muscles. Oropharyngeal exercise can be done with some facial movements .
  Arms: Oropharyngeal exercises

SUMMARY:
The effects of orofarangeal exercises (OE) and inspiratory muscle training (IMT) on sleep quality, disease severity, and airway muscle tone have been investigated in several studies. IMT and OE exercise modalities for patients and practitioners have advantages and disadvantages. It is recommended to compare exercise modalities in the studies. Whether OE or IMT exercise type is more effective on disease severity, sleep quality and snoring has not been investigated. The aim of this study was to compare the effectiveness of inspiratory muscle training and oropharyngeal exercises in patients with OSAS in terms of disease severity, snoring, daytime sleepiness, respiratory muscle strength and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

*To be diagnosed with mild, moderate and severe OSAS.

Exclusion Criteria:

* Patients with a history of stroke,
* neurological disease,
* severe obstructive nasal disease,
* and infection in the last month,
* BMI being 40 kg /m2 or more.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Polysomnography | 2 day
  Sleep efficiency, apnea-hypopnea index (AHI). Higher sleep efficiency and lower AHI values shows that patient have better status and lower disease severity

SECONDARY OUTCOMES:
Maximal inspiratory and expiratory muscle strength measurement with mouth pressure device | 6 day
  Respiratory muscle strength
6 minute walk test | 2 day
  Exercise capacity
Epworth Sleepiness Scale | 2 day
  minimum and maximum scores: 0-24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'
Berlin Questionnaire | 2 day
  Snoring frequency (0-3) and severity (0-4). Higher scores show higher snoring frequency and severity
Functional Outcomes of Sleep Questionnaire | 2 day
  Quality of life related with sleep. Minimum and maximum scores: 0-16. Higher scores show worse sleep related quality of life
The Pittsburgh Sleep Quality Index | 2 day
  Sleep quality. Minimum and maximum scores: 0-21. Higher scores show worse sleep quality
Fatigue Severity Scale | 2 day
  Fatigue severity. Minimum and maximum scores: 0-7. Scores higher than 4 shows high intensity fatigue perception

CONTACTS AND LOCATIONS:
Overall Officials: Adem Celik, MD, Study Chair — Ahi Evren Thoracic and Cardiovascular Surgery Hospital
Locations (1):
- Trabzon Ahi Evren Thoracic and Cardiovascular Surgery Training and Research Hospital, Trabzon, Turkey (Türkiye)